CLINICAL TRIAL: NCT05059704
Title: Effects of Circuit Class Training vs. Individual, Task Specific Training on Upper Extremity Function in Chronic Stroke Patient
Brief Title: Circuit Class Training vs. Individual, Task Specific Training in Chronic Stroke Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01036 Farwa Azmat
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Stroke
Keywords: Spasticity; Motor function
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Circuit Class Training (Experimental): Patients will participate in a total of 1.5hour/day for 8 weeks with a 1:3 (therapist to patient). The circuit will be divided into 5 specific stations, 5 to 10 minutes for warm-up tasks and 15 to 20 minutes on each station as tailored to the patient's activity level
  Interventions: Other: Circuit Class Training
- Individual Task specific training (Active Comparator): Patients will participate in a total of 1.5hour/day for 8 weeks with 1:1 (therapist to patient) ratio. During each session, all patients will perform 5 to 10 minutes warm-up tasks, then practiced the selected tasks for the rest of the time.
  Interventions: Other: Individual Task specific training

INTERVENTIONS:
Other: Circuit Class Training — Station 1 will include tasks for warm-up specific for upper extremity, station 2 will include shoulder exercises, station 3 will include elbow exercises, station 4 will include wrist exercises and station 5 will include hand activities and functional training. Variables such as speed, or/and resistance will progressively increase in diﬃculty according to each patient's ability.
  Arms: Circuit Class Training
Other: Individual Task specific training — Variables such as speed, or/and resistance will progressively increase in diﬃculty according to each patient's ability.
  Arms: Individual Task specific training

SUMMARY:
Due to minimal volitional activation of the impaired arm, these individuals are less able to engage in activities of daily living (ADL's). Moreover, simultaneous use of the hand and arm are needed throughout ADL's. The effects of these two approaches (circuit class training and individual task-specific training) on upper extremity function and activities of daily living (ADL's) have not yet been clearly identified, and studies on its effects on chronic stroke patients are limited.

DETAILED DESCRIPTION:
several research found that circuit training improved various functional parameters after stroke. And most of the circuit based tasks from the published studies were focused on the leg strength, walking speed, distance and balance etc. Previous literature found that circuit class training is effective in improving upper extremity function in chronic stroke patients disregarding the type of stroke and the results of that study are not generalized for chronic stroke patients with upper extremity deficit. Secondly, circuit class training and task-specific training are effective for improving upper limb function following a stroke but in the acute stage. In fact, there is no evidence in which comparison of these two approaches has been done in chronic stroke patients and thirdly, between these two approaches which approach is more effective towards improving upper limb function in chronic stage.

ELIGIBILITY:
Inclusion Criteria:

* Mini-Mental State Examination score more than 24
* Chronic stage (i.e. post-stroke duration of 6 months)
* Single episode of stroke
* MAS of 1 to 3 at upper extremity.
* MRS of ≤ 3 at lower extremity.
* MCA stroke
* Scores 32 to 47 on Fugl-Meyer Upper Extremity Scale (FMA-UE)

Exclusion Criteria:

* Orthopedic conditions that affect the UE function.
* Other neurological conditions, like PD, MS etc.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-06-26 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Scale | 8 weeks
  The Fugl-Meyer Assessment is the gold standard to assess motor function of post-stroke hemiparesis. The Fugl-Meyer Upper Extremity (FMUE) Scale is a widely used and highly recommended stroke-speciﬁc, performance-based measure of impairment. It is designed to assess reﬂex activity, movement control and muscle strength in the upper extremity of people with post-stroke hemiplegia.

SECONDARY OUTCOMES:
Modified Ashworth Scale | 8 weeks
  The modified Ashworth scale is the most universally accepted clinical tool used to measure the increase of muscle tone. The modified Ashworth scale is a muscle tone assessment scale used to assess the resistance experienced during passive range of motion, which does not require any instrumentation and is quick to perform
Stroke Specific-Quality of Life Urdu Version (SS-QOL) | 8 weeks
  The SS-QOL scale is a health-related outcome measure that comprises 49 items in 12 areas of vision, mobility, thinking, social roles, self-care, language, personality, family roles, work/productivity, upper limb function, mood and energy. It covers a more extensive inclusion of capacities ordinarily influenced by stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT(NMR), Principal Investigator — Riphah International University
Locations (1):
- Al Mustafa Trust Medical and Physiotherapy Centre, Dhok Gujra, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No